CLINICAL TRIAL: NCT01658319
Title: Phase I Trial of Fludarabine and Methoxyamine (TRC102) for Relapsed or Refractory Hematologic Malignancies
Brief Title: Methoxyamine and Fludarabine Phosphate in Treating Patients With Relapsed or Refractory Hematologic Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE2Y10; NCI-2010-02141 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2012-07-26; First posted 2012-08-07 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-08

CONDITIONS: Adult Nasal Type Extranodal NK/T-cell Lymphoma; Anaplastic Large Cell Lymphoma; Angioimmunoblastic T-cell Lymphoma; Cutaneous B-cell Non-Hodgkin Lymphoma; Extranodal Marginal Zone B-cell Lymphoma of Mucosa-associated Lymphoid Tissue; Hepatosplenic T-cell Lymphoma; Intraocular Lymphoma; Nodal Marginal Zone B-cell Lymphoma; Peripheral T-cell Lymphoma; Recurrent Adult Burkitt Lymphoma; Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Adult Diffuse Mixed Cell Lymphoma; Recurrent Adult Diffuse Small Cleaved Cell Lymphoma; Recurrent Adult Grade III Lymphomatoid Granulomatosis; Recurrent Adult Hodgkin Lymphoma; Recurrent Adult Immunoblastic Large Cell Lymphoma; Recurrent Adult Lymphoblastic Lymphoma; Recurrent Adult T-cell Leukemia/Lymphoma; Recurrent Cutaneous T-cell Non-Hodgkin Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Marginal Zone Lymphoma; Recurrent Mycosis Fungoides/Sezary Syndrome; Recurrent Small Lymphocytic Lymphoma; Refractory Chronic Lymphocytic Leukemia; Refractory Multiple Myeloma; Relapsing Chronic Myelogenous Leukemia; Small Intestine Lymphoma; Splenic Marginal Zone Lymphoma; Stage III Chronic Lymphocytic Leukemia; Testicular Lymphoma; Waldenström Macroglobulinemia
MeSH Terms: conditions — Lymphoma, Extranodal NK-T-Cell; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Intraocular Lymphoma; Lymphoma, B-Cell, Marginal Zone; Lymphoma, T-Cell, Peripheral; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Hodgkin Disease; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Mycosis Fungoides; Sezary Syndrome; Leukemia, Lymphocytic, Chronic, B-Cell; Multiple Myeloma; Waldenstrom Macroglobulinemia | interventions — fludarabine phosphate; methoxyamine; Blotting, Western; Mass Spectrometry

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (chemotherapy) (Experimental): Patients receive fludarabine phosphate IV over 30 minutes on days 1-5 and methoxyamine IV over 1 hour on day 1 (day 2 of course 1). Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: fludarabine phosphate; Drug: methoxyamine; Other: laboratory biomarker analysis; Other: pharmacological study; Genetic: western blotting; Other: mass spectrometry; Genetic: DNA analysis

INTERVENTIONS:
Drug: fludarabine phosphate — Given IV
  Other Names: 2-F-ara-AMP; Beneflur; Fludara
Drug: methoxyamine — Given IV
  Other Names: TRC102
Other: laboratory biomarker analysis — Correlative studies
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Genetic: western blotting — Correlative studies
  Other Names: Blotting, Western; Western Blot
Other: mass spectrometry — Correlative studies
Genetic: DNA analysis — Correlative studies

SUMMARY:
This phase I trial is studying the side effects and best dose of methoxyamine when given together with fludarabine phosphate in treating patients with relapsed or refractory hematologic malignancies. Drugs used in chemotherapy, such as methoxyamine and fludarabine phosphate, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving methoxyamine together with fludarabine phosphate may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) of methoxyamine given in conjunction with fludarabine (fludarabine phosphate) in subjects with relapsed or refractory hematologic malignancies.

SECONDARY OBJECTIVES:

I. To determine the dose limiting toxicities of the combination of methoxyamine and fludarabine.

II. To determine the pharmacokinetics of methoxyamine when given in combination with fludarabine.

III. To evaluate pharmacodynamic endpoints including apurinic/apyrimidinic (AP) sites and deoxyribonucleic acid (DNA) strand breaks in blood mononuclear cells to explore the in vivo mechanism of action of methoxyamine and identify the biologically optimal dose to be combined with fludarabine.

VI. To determine the disease specific toxicity and biologic activity in a cohort of chronic lymphocytic leukemia (CLL) patients.

OUTLINE: This is a dose-escalation study of methoxyamine.

Patients receive fludarabine phosphate intravenously (IV) over 30 minutes on days 1-5 and methoxyamine IV over 1 hour on day 1 (day 2 of course 1). Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have a histologically confirmed hematologic malignancy that has relapsed or proven refractory (in any time frame) to one or more prior therapies, limited to the following subtypes:

  * Non-Hodgkin lymphoma (NHL), including cutaneous lymphoma
  * Hodgkin lymphoma (HL)
  * Chronic lymphocytic leukemia (CLL)
  * Chronic myeloid leukemia (CML)
  * Multiple myeloma
* Patients must have progressed through standard curative treatment options in the case of NHL and HL or not be candidates for curative therapy
* Patients must have measurable disease, and must meet criteria justifying a need to initiate therapy, criteria for measurable disease and criteria for initiating therapy for purposes of this study are defined as follows:
* NHL/HL: measurable disease by radiographic criteria (>= 1 cm by computed tomography); or any degree of bone marrow involvement with lymphoma by morphologic analysis; or measurable skin involvement according to cutaneous lymphoma response criteria; criteria for initiating therapy include aggressive histology (diffuse large B cell lymphoma, nodal T cell lymphomas, Hodgkin lymphoma) or presence of any of the following: systemic symptoms, bulk >= 5 cm, >= 3 nodal sites, marrow compromise remaining within limits of adequate function as defined below, splenomegaly >= 16 cm, disease-related effusion, risk of local compressive symptoms, or circulating lymphoma cells
* CLL: measurable disease requires B lymphocytes equal or greater than 5,000/μL, or lymphadenopathy (>= 1 cm by computed tomography), or bone marrow involvement of any degree; in addition, patients must have one of the following: Rai stage III (hemoglobin < 11gm/dL) or IV (platelets < 100,000/uL) disease, progressive splenomegaly, hepatomegaly or lymphadenopathy, weight loss > 10% over the preceding 6 month period, grade 2 or 3 fatigue, fevers > 100.5 or night sweats without evidence for infection, progressive lymphocytosis with an increase of > 50% over a 2 month period or an anticipated doubling time of < 6 months
* Chronic Myeloid Leukemia: measurable disease requires peripheral or bone marrow evidence of CML by hematologic, cytogenetic, or molecular analysis; any patient meets criteria for initiating therapy who has failed >= 1 prior treatment with a tyrosine kinase inhibitor (relapsed or refractory)
* Multiple myeloma: measurable disease and presence of end-organ damage; measurable disease includes any of the following: abnormal free light chain (FLC) ratio, an M-component in the serum or urine, clonal plasma cells in the bone marrow and/or a documented clonal plasmacytoma; end-organ damage includes any of the following: calcium elevation (> 11.5 mg/dl), anemia (hemoglobin < 10 g/dl), bone disease (lytic lesions or osteopenia), or renal involvement (proteinuria or any known nephropathy) as long as Cr < 1.5 mg/dL
* Prior chemotherapy and/or radiation are allowed; at least 3 weeks must have elapsed since prior large-field radiation therapy; patients must have been off previous anti-cancer therapy for at least 3 weeks. Non - hematologic acute treatment related toxicities must have resolved to a grade 2 or less, whereas non hematologic chronic treatment related toxicities must be stable or shown improvement in the 4 weeks preceding enrollment. Because of the nature of the diseases treated in this protocol, hematologic toxicities are not included in this criterion and must meet the eligibility criteria described above. At least 12 weeks must have passed since radioimmunotherapy; prior fludarabine treatment is not restricted
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Life expectancy > 12 weeks
* Absolute neutrophil count > 750/ul
* Platelets > 50,000/ul
* Hemoglobin > 9.0 g/dl
* Total bilirubin < 1.5 mg/dl
* Aspartate aminotransferase (AST)(serum glutamic oxaloacetic transaminase [SGOT]) < 2.5 x institutional upper limit of normal
* Creatinine < 1.5 mg/dl and/or creatinine clearance > 60 mL/min/1.73 m^2
* Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients may not be receiving any other investigational agents or have received other investigational agents for at least 3 weeks
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant and lactating women are excluded from this study
* New York Heart Association (NYHA) classification III or IV heart disease
* Uncontrolled brain or leptomeningeal metastases, including patients who continue to require glucocorticoids for brain or leptomeningeal metastases
* Known seizure disorder
* Known human immunodeficiency virus (HIV) or chronic hepatitis (B or C) infection
* Patients unwilling or unable for any reason (personal, medical, or psychiatric) to comply with the protocol
* Patients with known hypersensitivity to fludarabine or a history of purine analog associated autoimmune hemolytic anemia or idiopathic thrombocytopenic purpura

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-05; Primary Completion 2015-02 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of methoxyamine given in conjunction with fludarabine in subjects with relapsed or refractory hematologic malignancies | one cycle (28 days)
  Defined as the highest dose tested in which none or only one subject experiences a dose limiting toxicities attributable to the study drug combination during the first cycle of treatment, when 3-6 subjects were treated at that dose and are evaluable for toxicity.
MTD of methoxyamine given in conjunction with fludarabine in subjects with relapsed or refractory hematologic malignancies | after 6 cycles (at 6 months)
  Defined as the highest dose tested in which none or only one subject experiences a dose limiting toxicities attributable to the study drug combination during the first cycle of treatment, when 3-6 subjects were treated at that dose and are evaluable for toxicity.

SECONDARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Dose limiting toxicities of the combination of methoxyamine and fludarabine | at 6 cycles (6 months) of treatment
Number of Participants with Adverse Events as a Measure of Dose limiting toxicities of the combination of methoxyamine and fludarabine | 1 year
Pharmacokinetics of methoxyamine when given in combination with fludarabine as determined by methoxyamine levels at different time points. | On day 2, immediately before and 2 hours after the initialmethoxyamine treatment, on days 3-5, and when the patient returns for fludarabine administration and on day 8
  The estimated total dose of methoxyamine given over a 60 minute i.v. infusion needed to produce a Cmax of 41.40 ng/mL (60.40 mg) corresponds to 30 mg/m2 (assuming an average BSA of 2 m2), representing a rational and safe starting methoxyamine dose to administer intravenously over 60 minutes.
Number of apurinic/pyrimidinic (AP) sites. | At 0, 2, 24, 27, 48, 72 and 96 hours post fludarabine-treatment
  Use aldehyde reactive probe (ARP) reagent to measure AP sites formed by fludarabine and blocked by methoxyamine. AP sites will be measured on DNA extracted from patients' mononuclear cells. Analysis of AP site and DNA strand breakage will be used to determine the biologically optimal dose of methoxyamine to be used in combination with fludarabine.
Change in miRNA profiles in CLL cells in a cohort of CLL patients | Baseline and at 2hrs and 27 hours after treatment
  Specific microRNA (miRNA) expression patterns will uniquely predict the clinical response of CLL patients after exposure to Fludarabine alone or in combination with Methoxyamine (MX) in this phase I clinical trial.
Number of DNA strand breaks determination by comet assay to monitor drug effects on DNA damage in clinical studies. | At 0, 2, 24, 27, 48, 72 and 96 hours post fludarabine-treatment
  Analysis of AP site and DNA strand breakage will be used to determine the biologically optimal dose of methoxyamine to be used in combination with fludarabine.
Measure of Proteins (Bcl-2, Bax, cleaved PARP, Topoisomerase I and II, GammaH2AX) | day 0h (day1), at 24h (day2) and 48h (day3) prior to drug injection at each time point
  Results of the protein assays will be used to further elucidate how methoxyamine potentiates fludarabine induced apoptosis and to evaluate potential synergy between the 2 agents.

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Caimi, MD, Principal Investigator — Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center
Locations (1):
- Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States